CLINICAL TRIAL: NCT05303207
Title: Study to Evaluate the Efficacy of YOUR SUPER Detox Bundle to Improve Perceived Well Being and Promote Adaptation of Healthy Dietary Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Your Super, INC. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20233YourSuper
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Eating Habit; Healthy Diet
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Your Super Detox (Other): Dietary supplement
  Interventions: Dietary Supplement: YOUR SUPER Detox Bundle

INTERVENTIONS:
Dietary Supplement: YOUR SUPER Detox Bundle — During days 1-5, participants will complete the 5-day Your Super Detox, consuming 2 smoothies daily (breakfast and dinner) containing Your Super Detox superfood powders.

SUMMARY:
This is an open-label observational single-group clinical trial to study the efficacy of a commercial superfood blend and its effect on markers of well-being and improvement of long-term healthy eating habits.

DETAILED DESCRIPTION:
This is an open-label observational single-group clinical trial to study the efficacy of a commercial superfood blend and its effect on markers of well-being and improvement of long-term healthy eating habits.

It is hypothesized that the dietary supplement marketed as Your Super Detox Bundle will improve subjective wellbeing and health in trial participants. It is further hypothesized that the accompanying diet plan will promote beneficial nutritional habits that may persist long term outside of the 5-day detox period. Additionally, the included food ingredients are reported to improve energy levels and sleep quality, while reducing unfavorable bloating, aches, and brain fog.

A total of 38 participants will be recruited for the trial following the screening. The trial will be fully remote, a technology platform will be utilized to screen, enroll and capture study data of the participants. Participants will undergo a 5-day detox period involving consuming two smoothies daily (for breakfast and dinner) containing variations of the Your Super Detox food powders as detailed below. Participants are encouraged to follow the provided plant-based nutritional plan for meals and snacks outside of the Your Super smoothie meals. Participant adherence to the provided nutritional plan is not mandatory, and lack of adherence by some participants will provide further data on the effect of the nutritional guidelines on the evaluated outcomes. After the 5-day detox period is completed, participants will be followed on for a subsequent 16 days to evaluate the effect of Your Super Detox bundle and guidelines to influence prolonged healthy eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Male & Female
* Age 18-55
* Feeling fatigued often
* Eating fast food, such as fries, burgers, pizza, chicken wings, etc. at least twice a week
* Does not exercise regularly
* Does not consume fruits and vegetables regularly
* Must be in generally good health - no unstable, uncontrolled health condition
* BMI under 40
* May feel bloated often
* May experience gas production often
* May experience heartburn
* May experience irritable bowel symptoms
* May experience irregular bowel movements
* May experience regular body aches
* May experience regular joint, back or neck pain
* Must have a body scale at home for regular weigh-in

Exclusion Criteria:

* Severe chronic conditions, including oncological and psychiatric disorders
* Known to have any severe allergic reactions
* Currently pregnant, breastfeeding, or wanting to become pregnant for the duration of the study
* Participants unwilling to follow the study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in perceived commitment to long-term healthy eating habits | 5 days
  The study uses a questionnaire to assess the effectiveness of the intervention on a scale from 0-5 (0=Lowest score and 5=Highest score).

SECONDARY OUTCOMES:
Changes in well-being markers of well being | 5 days
  The study uses a questionnaire to assess changes in well-being on a scale from 0-5 (0=Lowest score and 5=Highest score).

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No